CLINICAL TRIAL: NCT05492799
Title: Open-Label Multicenter Extension Study to Further Evaluate Safety, Tolerability and Efficacy of Intracerebroventricular AX 250 Treatment in Mucopolysaccharidosis Type IIIB (MPS IIIB, Sanfilippo Syndrome Type B) Patients
Brief Title: Safety, Tolerability and Efficacy of ICV AX 250 Treatment in MPS IIIB -OLE
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Allievex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250-401
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: MPS III B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): AX 250 300 mg - open label
  Interventions: Drug: AX 250

INTERVENTIONS:
Drug: AX 250 — biweekly infusion by intracerebroventricular (ICV) infusion

SUMMARY:
This is a Phase 3B/4, multicenter, multinational, open label study to further evaluate intracerebroventricular (ICV) delivered AX 250 treatment in MPS IIIB subjects that complete Study 250-202 for up to an additional 3 years (144 weeks) of treatment with AX 250 administered by ICV infusion every other week. Subjects will be evaluated for neurocognitive function, communication, adaptive behavior, quality of life, imaging characteristics and biochemical markers of disease burden. Safety will be assessed by adverse events, clinical labs, and physical exams.

ELIGIBILITY:
Inclusion Criteria:

1. Must have completed 240 weeks of Study 250-202 and enter 250-401 within 8 weeks of dosing completion.
2. Provides written informed consent from parent or legal guardian and assent from subject, if required
3. Has the ability to comply with protocol requirements in the opinion of the investigator
4. If female with childbearing potential, must have a negative pregnancy test at the Screening visit and be willing to have additional pregnancy tests during the study

Exclusion Criteria:

1. Has (1) a cognitive age equivalent (AEq ) score ≤ 18 months, (2) a development quotient (DQ) score ≤ 20, and (3) no evidence of improvement during the 250-202 study in secondary or exploratory efficacy endpoints
2. Would not benefit from enrolling in the study in the opinion of the investigator
3. Has received stem cell, gene therapy or enzyme replacement therapy (other than AX 250) for MPS IIIB
4. Has a history of poorly controlled seizure disorder
5. Is prone to complications from ICV drug administration including patients with hydrocephalus or ventricular shunts
6. Has received any investigational medication within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
7. Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's well-being or safety, or the interpretability of the subject's clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary - neurocognition | baseline to 144 weeks of treatment
  the rate of change in score from neurocognitive assessment using validated scale

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allievex Corporation
Locations (6):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UPMC Children's Hospital Pittburgh, Pittsburgh, Pennsylvania
- Fundación Cardio Infantil - Instituto de Cardiología, Bogotá, Colombia
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Great Ormond Street Hospital For Children, NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No